CLINICAL TRIAL: NCT05191407
Title: Investigation of Factors Associated With the Increased Fear and Anxiety in Dental Patients During the COVID-19 Pandemic in Turkey: A Survey
Brief Title: Fear and Anxiety Level in Dental Patients During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Zeliha Aytekin (Other)
Responsible Party: Sponsor-Investigator, Zeliha Aytekin, Research Assistant, Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: 70904504 /706
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Fear; Anxiety; COVID-19
Keywords: COVID-19 Pandemic; COVID-19; fear; anxiety
MeSH Terms: conditions — Anxiety Disorders; COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Biological samples were not taken from individuals in the study. The study is a survey study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psychological support may be needed to help patients in the face of emotional disturbances that may be associated with the outbreak and to help them accomplish their fear and anxiety. Due to the increasing fear of COVID-19 transmission during the pandemic, patients may develop treatment avoidance behavior in dental practices. If the fear and anxiety levels of the patients can be determined, it may be easy to offer special approaches to them.

DETAILED DESCRIPTION:
Officially, the first COVID-19 case in Turkey was diagnosed on March 10, 2020. To ensure social isolation, cities were locked down with residents to stay at home to prevent disease transmission. A very large part of the population may experience frustration, stress, and irritability while in isolation. Due to the prolonged lockdown and COVID-19 associated fear, the COVID-19 pandemic, which threatens people's physical health and lives, is likely to trigger a wide variety of psychological problems such as anxiety and depression by increasing their stress levels.

The risk of cross-infection in dentistry has been described as considerably high due to close physical contact between dental professionals and patients, and aerosols production during routine dental treatments. In this uncertain process, patients remain undecided about attending their dental appointments. Their concern is associated with the risk of getting infected and transmitting the disease to family members. All these factors may increase the mental stress of patients.

The essential purpose of this study is to evaluate the COVID-19 fear and anxiety level, COVID-19 knowledge status, and information sources in dental patients in Turkey during the pandemic period.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate with providing informed consent;
* age ≥18 years
* able to understand and read & write the Turkish language.

Exclusion Criteria:

* not willing to participate with providing informed consent;
* age<18 years
* not able to understand and read & write the Turkish language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals randomly selected from the patients who applied to the Faculty of Dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
fear of COVID-19 | last six month ( from the beggining of the pandemic to time of survey)
  The fear of participants is measured by the Turkish validated version of the fear of COVID-19 Scale.
anxiety | last two weeks
  The anxiety level of the participants is measured by the Turkish version of Generalized Anxiety Disorder-7 Scale

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Daltaban, PhD, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Temsah MH, Al-Sohime F, Alamro N, Al-Eyadhy A, Al-Hasan K, Jamal A, Al-Maglouth I, Aljamaan F, Al Amri M, Barry M, Al-Subaie S, Somily AM. The psychological impact of COVID-19 pandemic on health care workers in a MERS-CoV endemic country. J Infect Public Health. 2020 Jun;13(6):877-882. doi: 10.1016/j.jiph.2020.05.021. Epub 2020 May 29. PMID 32505461
- [Result] Al-Rahimi JS, Nass NM, Hassoubah SA, Wazqar DY, Alamoudi SA. Levels and predictors of fear and health anxiety during the current outbreak of COVID-19 in immunocompromised and chronic disease patients in Saudi Arabia: A cross-sectional correlational study. PLoS One. 2021 Apr 26;16(4):e0250554. doi: 10.1371/journal.pone.0250554. eCollection 2021. PMID 33901260